CLINICAL TRIAL: NCT06422871
Title: PReSeRVE-HD: PRospective, Multicenter, Observational Study of the Merit HeRO® Graft and Super HeRO® EValuated in End-Stage Renal Disease Patients on HemoDialysis
Brief Title: PReSeRVE-HD: Observational Study of the Merit HeRO® Graft and Super HeRO® in Patients on Hemodialysis
Acronym: PReSeRVE-HD
Status: Recruiting | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CVO-P4-23-02
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: End Stage Renal Disease; Hemodialysis Access Failure
Keywords: HeRO
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- HeRO® / Super HeRO®: Subjects who meet all inclusion criteria and none of the exclusion criteria and treatment is attempted with the HeRO® Graft or Super HeRO® device.
  Interventions: Device: HeRO® Graft System or Super HeRO® System

INTERVENTIONS:
Device: HeRO® Graft System or Super HeRO® System — Treatment attempted with the HeRO® or Super HeRO® device.

SUMMARY:
The goal of this observational study is to increase the understanding of the safety and performance of Merit Medical's HeRO Graft System (HeRO) and Super HeRO Adaptor and Support Seal System (Super HeRO) devices. This study includes adults that are being treated with one of these devices as part of their regular medical care for maintaining long-term dialysis access when all other dialysis access options have failed. If participants in the study are not seen for a standard of care clinic visit during the 4 visit timepoints over 2 years, the participant will be followed by phone to check their current health and dialysis status.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject provides written informed consent
* Subject is ≥ 18 years
* Subject is end-stage renal disease patient on hemodialysis.
* Subject is treated with HeRO Graft or Super HeRO System in accordance with device instructions for use (IFU)

Key Exclusion Criteria:

* Subject has a previously placed HeRO or Super HeRO device that is undergoing revision or replacement
* Subject has a topical or subcutaneous infection associated with the implantation site
* Subject has known or suspected systemic infection, bacteremia or septicemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients on hemodialysis who have exhausted all other access options.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint | 6 months
  Clinical Success, defined as maintenance of access circuit patency in the absence of device-related infection or bacteremia

SECONDARY OUTCOMES:
Clinical Success | 12 and 24 months
Proportion of subjects with primary patency | 6, 12 and 24 months
Proportion of subjects with cumulative patency | 6, 12, and 24 months
Device-related safety events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hohmann, MD, Principal Investigator — Baylor Scott and White Health
Locations (3):
- United States (3):
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - WakeMed, Raleigh, North Carolina
  - Baylor Scott & White Heart and Vascular Hospital - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No